CLINICAL TRIAL: NCT03045978
Title: The Role of Ghrelin, Leptin, Adiponectin, Neuropeptide Y, Orexin A, Insulin Like Growth Factor-1(IGF-1), IGFBP-1, IGFBP-3, Corticotrophin-releasing Hormone in Feeding and Nutritional Consequences in Children With Feeding Difficulty.
Brief Title: The Association of Hormones and Peptides With Nutritional Consequences in Children With Feeding Difficulty.
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 103-7090A3
Record Dates: First submitted 2017-01-13; First posted 2017-02-08 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2017-01

CONDITIONS: Feeding Difficulty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood is collected in Serum separation tubes and kept at 4 °C for 1 before being centrifuged, and the serum is stored at -80 °C.
Oversight: Data Monitoring Committee: No

SUMMARY:
To study the role of ghrelin, leptin, adiponectin, neuropeptide Y (NPY), orexin A, IGF-1, IGFBP-1, IGFBP-3, and corticotrophin-releasing hormone (CRH) in the nutritional status in children with feeding difficulty, and further to evaluate their regulation with feeding difficulties (anorexia, picky eating behavior, feeding disorders with concurrent medical conditions).

DETAILED DESCRIPTION:
The investigations plan to prospectively evaluate the plasma concentration of endocrine parameters in children with feeding difficulties. The studied children are arranged to do the dietary records, clinical survey and laboratory studies at the inpatient or outpatient department at clinical evaluation and follow-up. The duration of evaluation and follow-up is 3 months. The healthy children in the control group are also assigned to do the dietary records, clinical survey and laboratory studies after exclusion of feeding difficulty and malnutrition by feeding and nutritional assessment (same survey as the studied patients demonstrated in the following section "clinical survey"). The healthy children do not need the follow-up assessment at 12 weeks.

The diagnosis of feeding difficulty is based on "IMFeD" program. The categorizations of feeding difficulties in the IMFeD tool was originally developed by Dr. Chatoor and Dr. Kerzner (Clinical investigation of feeding difficulties in young children: a practical approach, Clinical Pediatrics, 2009). The 7-day dietary records and assessment of daily calories are evaluated by dietician and research assistant. Nutritional assessment includes 7-day dietary record, assessment of daily calories, body weight (BW), body height (BH), weight for age z-score, height for age z-score, BMI, BMI for age z-score, weight for height index, weight-for-height z-score, severity of malnutrition, and nutritional serum markers (hemoglobin, lymphocyte count, pre-albumin, albumin, ferritin, and zinc). Growth standards for height, weight, and BMI based on World Health Organization (WHO) population were used to obtain z-scores for each measurement, according to age and gender. The severity of malnutrition is determined by weight-for-height.

The laboratory studies will be performed at baseline and at 12 weeks. Venous blood is collected in Serum separation tubes and kept at 4 °C for 1 before being centrifuged, and the serum is stored at -80 °C. All measurements are performed in the same assay without extraction. Concentrations of serum ghrelin, leptin, adiponectin, NPY, orexin A, IGF-1, IGFBP-1, IGFBP-3 and CRH are all determined using enzyme-linked immunosorbent assay (ELISA) kits. All assays were performed according to the manufacturers' instructions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with feeding difficulties are evaluated by the children gastroenterologist. The diagnosis of feeding difficulty is based on "IMFeD" program.
2. Children aged 2-18 years old with feeding difficulty are enrolled.

Exclusion Criteria:

1. pernicious anemia
2. dysfunction of blood coagulation
3. leukemias
4. infection in skin of the blood collection sites
5. edema, poor circulation or severe trauma of limb
6. phlebitis or vein thrombosis

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1. Studied subjects: children with clinical diagnosis of feeding difficulty.
  2. Methods of study: A total of 90 children aged 2-12 years old with feeding difficulty are enrolled into the study, and 30 healthy children are used as control. The enrolled subjects with feeding difficulty are assigned clinical survey for 12 weeks and laboratory studies at enrollment and at 12 weeks, and they are classified into 3 groups: (1) Group 1: 30 patients without malnutrition, (2) Group 2: 30 patients with mild malnutrition, and (3) Group 3: 30 patients with marked malnutrition.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The change of hormones and growth factors levels in laboratory data | Changes from baseline to week 12.
  Observe the level of ghrelin, leptin, adiponectin, Neuropeptide Y, orexin A, Insulin-like growth factor 1, insulin-like growth factor-binding protein 1, insulin-like growth factor-binding protein 3 and corticotropin-releasing hormone in the laboratory data.

CONTACTS AND LOCATIONS:
Overall Officials: Hsun-Chin Chao, A.P., Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No